CLINICAL TRIAL: NCT00166556
Title: Thistlethwaite Protocol # ITN025ST - Immunosuppression With Campath-1H and Tacrolimus in Liver Transplantation
Brief Title: A Trial to Assess Campath-1H and Tacrolimus Followed by Immunosuppression Withdrawal in Liver Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: University of Chicago (Other); Immune Tolerance Network (ITN) (Network)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2355-04
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2011-05-23 (Estimated); Status verified 2011-05

CONDITIONS: Transplantation, Liver
MeSH Terms: interventions — Alemtuzumab; Tacrolimus

INTERVENTIONS:
Drug: Campath-1H and Tacrolimus

SUMMARY:
This is a prospective, multicenter open-label single arm trial in which recipients of liver allograft will receive uniform immunosuppressive induction and maintenance regimens. Participants with end stage liver disease who meets the entry criteria will be consented and enrolled.

Participants receive Campath-1H and maintenance immunosuppression with tacrolimus therapy. After one year of tacrolimus therapy, an assessment of the immunologic status including blood gene expression and geno-race studies will be performed which will include studies on the liver graft biopsy. At this time, patients will be selected to undergo immunosuppressive withdrawal. This will be made on an individual basis with definitive inclusion and exclusion criteria.

The objectives of the study are to evaluate the safety and efficacy of immunosuppressive regimens comprising Campath-1H induction followed by maintenance immunosuppressive therapy with tacrolimus on allograft survival. However, secondary objectives will be to assess withdrawing tacrolimus after Campath-1H induction in an immune depletion and subsequent immune reconstitution. This study will evaluate whether a combination of anti-rejection medications (Campath-1H and tacrolimus) can prevent rejection and allow the body to develop tolerance to the transplanted liver.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18 years of age or older
2. Necessity for liver transplant
3. A negative pregnancy test at study entry for females of child-bearing potential
4. For participants with reproductive potential, agreement to use approved methods of birth control for the duration of their participation
5. Ability to provide informed consent
6. Availability of donor spleen

Exclusion Criteria:

1. Previous transplant
2. Multiorgan transplant
3. Living donor transplant.
4. Donor liver from a donor positive for antibody against hepatitis B core antigen
5. Donor liver from a donor positive for antibody against hepatitis C
6. Donor liver from a non-heart-beating donor
7. Liver failure due to autoimmune disease, such as autoimmune hepatitis, primary sclerosing cholangitis, and primary biliary cirrhosis
8. Hepatitis B infection as defined by the presence of HbSAg or active treatment for hepatitis B
9. Hepatitis C as defined by the presence of antibody against hepatitis C.
10. Stage III or higher hepatocellular cancer based on pretransplant imaging
11. History of malignancy except hepatocellular cancer, or adequately treated in situ cervical carcinoma, adequately treated basal or squamous cell carcinoma of skin, or other malignancy which is judged to have a 5-year risk of recurrence of < 5%
12. Active systemic infection at the time of transplantation
13. Clinically significant chronic renal disease
14. Clinically significant cardiovascular or cerebrovascular disease
15. Infection with human immunodeficiency virus
16. Any investigational drug received within 6 weeks of study entry
17. Hypersensitivity to Campath-1H or tacrolimus
18. Unwillingness or inability to comply with study requirements (Immune Tolerance Network CONFIDENTIAL iv Protocol ITN024ST Immunosuppression with Campath-1H Version 3.0 June 28, 2005 and Tacrolimus in Liver Transplantation)
19. Inability to give appropriate informed consent (e.g., hepatic encephalopathy stage 2 or higher at time of screening consent)
20. Positive PPD without evidence of prior treatment or administration of BCG

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2005-01; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of an immunosuppression regimen comprising Campath-1H induction followed by maintenance therapy with tacrolimus in allowing liver allograft survival

SECONDARY OUTCOMES:
Assess the safety of withdrawing tacrolimus after Campath-1H induced immuno-depletion and subsequent immune reconstitution
Gather additional safety information about the combination of Campath-1H and tacrolimus in liver allograft recipients
Define profiles of immunologic and genetic features present prior to or during tapering of immunosuppression that distinguish tolerant and non tolerant allograft recipients

CONTACTS AND LOCATIONS:
Overall Officials: Russell H. Wiesner, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States